CLINICAL TRIAL: NCT04705792
Title: Physical Rehabilitation in Adults With Sickle Cell Anemia: Effects on Muscle Function, Functional Capacity and Quality of Life
Brief Title: Physical Rehabilitation in Sickle Cell Anemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.718.917/2016
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Sickle Cell Anemia; Muscle Dysfunction; Quality of Life; Physical Activity; Exercise
Keywords: Sickle Cell Anemia; Rehabilitation; Physiotherapy
MeSH Terms: conditions — Anemia, Sickle Cell; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: After a physical therapy evaluation, the patient underwent a booklet-guided physical exercise program that lasted three months (3 times per week with a duration of 60 minutes per session). Activities included overall stretching and strengthening (flexion, extension, adduction and abduction movements) and muscular endurance exercises (exercises involving open and closed kinetic chains), along with aerobic conditioning using a functional circuit. The patient was evaluated at 2 different timepoints (baseline and after 12 weeks of training); thus, he served as his own control. The physiotherapist contacted the patient by phone weekly to follow the progression of the treatment. Throughout the application of the protocol, the patient regularly maintained his follow-up visits with the multidisciplinary team. Moreover, there was no change in pharmacological treatment throughout this period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity (Experimental): The program comprises the practice of resistance exercises for the main muscular groups, with free weights and with their own body weight against the action of gravity, the proposal consists of 3 weekly sessions, for 12 consecutive weeks.
  Interventions: Procedure: Physical activity

INTERVENTIONS:
Procedure: Physical activity — Activities included overall stretching and strengthening (flexion, extension, adduction and abduction movements) and muscular endurance exercises (exercises involving open and closed kinetic chains), along with aerobic conditioning using a functional circuit.

SUMMARY:
Sickle cell anemia (SCA) is one of the most neglected diseases worldwide, according to the World Health Organization. In the adult population with SCA, the systemic effects of the disease, such as respiratory and peripheral muscle dysfunction, cause a decrease in quality of life. As a consequence, there is a concern about functional rehabilitation, since the aging of this population is already a reality in our environment. Thus, the objective of this project is to evaluate the effects of functional rehabilitation on quality of life in adult patients over 18 years of SCA. In this longitudinal intervention study, patients will be submitted to a three-month rehabilitation program. Before and after the intervention, patients will be submitted to the following assessments: spirometry; quality of life questionnaire - Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36); functional scale of joint integrity - Lower Extremity Functional Scale (LEFS); fatigue assessment scale - Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F); physical activity assessment questionnaire - International Physical Activity Questionaire (IPAQ); peripheral muscle assessment (handgrip and isometric dynamometry of the quadriceps muscle); and 6-minute walk test (6MWT). The protocol will consist of warm-up and cool-down exercises, muscle strengthening and endurance exercises, aerobic training, balance training and proprioception. Thus, it is expected that patients with sickle cell anemia will benefit significantly, with a consequent improvement in musculoskeletal function, pain and health-related quality of life.

DETAILED DESCRIPTION:
Over the past 40 years, Public Health measures have led to an impressive decline in infant mortality related to sickle cell disease (SCA) and, thus, modified its evolution. Sickle cell disease went from a life-threatening disease in childhood in the 1970s to a chronic disease of adults today. In Brazil, the median age of cases that evolved to death was 26.5 years in Bahia, 31.5 years in Rio de Janeiro and 30 years in São Paulo. In a study carried out in Minas Gerais, the average age at the time of death was 33.5 years considering only adults; this was higher in the female gender (46.5 years) and the majority occurred as a result of acute events.

Osteoarticular and muscle involvement is common in adults with sickle cell disease and has high morbidity. Since bone microcirculation is a place where sickling of red blood cells is common, there is a tendency for thrombosis, infarction and necrosis. The osteoarticular lesion is characterized mainly by osteonecrosis, osteomyelitis and arthritis, with frequent involvement of the hip and shoulder bones and the vertebral bodies.

Bone changes in SCA can be grouped into two main forms: those associated with ischemic events and those associated with bone marrow hyperplasia due to chronic anemia. The pathogenesis of microvascular occlusion, the key event of vaso-occlusive crises, is complex and involves the activation of leukocytes, platelets and endothelial cells, in addition to hemoglobin S containing red blood cells. These events can occur in almost any organ, but are particularly common in the bone marrow, possibly because of its hypercellularity, leading to a decrease in blood flow and regional hypoxia. There is also evidence of a possible association between changes in calcium metabolism and the occurrence of osteoporosis in people with sickle cell disease.

Regarding muscle disease, some studies have shown a decrease in both muscle strength and endurance in individuals with sickle cell disease. General amyotrophy results from repeated episodes of vasoocclusion and ischemia of the muscles, sometimes silent or subclinical, which occur in sickle cell anemia and are known to induce dysfunction and, eventually, skeletal muscle necrosis. Sickle cells and oxidative stress can cause microvascular obstruction and damage peripheral muscles in patients with SCA. Consequently, there are marked changes in skeletal muscle structure, with rarefaction of microvessels and decreased capillary tortuosity.

The main cause of emergency care for people with SCA is painful osteoarticular crises, which are observed in about 70% of cases, while the most frequent complications that require hospitalization in these individuals are the vaso-occlusive crisis and osteomyelitis. Other bone complications in acute SCA are stress fractures, orbital compression, vertebral collapse and spinal necrosis.

Osteonecrosis is a frequent complication in SCA, manifesting through painful and debilitating findings, and 50% of patients with the disease have evidence of complications after the age of 30. Spinal bone injury has been attributed to areas of bone infarction that can reach the central portions of the vertebral plateau and, as a consequence, lead to overgrowth of the adjacent portions and central depression of the plateau. Vaso-occlusive seizures mainly affect long bones, but they can also occur in the vertebrae and ribs and cause complications of respiratory function. Osteonecrosis of the femoral head has an incidence of 4.5 cases per 100 patients/year, often being bilateral. These vaso-occlusive crises are caused by obstructions in the microcirculation and are favored by some factors, such as prolonged immobilization, physical exercise, sudden changes in temperature, fever and dehydration.

Muscle weakness may be the result of the pathophysiology of SCA, in which patients have frequent vaso-occlusive crises due to the polymerization process of the hemoglobin S, which promotes greater adhesion of these cells to the vascular endothelium and can induce ischemia, inflammation and oxidative stress . It is known that oxidative stress can damage the peripheral muscles, causing damage to the performance of these muscles. The systemic damage caused by SCA can also lead to a more sedentary lifestyle, which, in turn, can result in an overall loss of muscle strength with a consequent reduction in functional capacity.

SCA is a chronic disease in which a cure is not yet possible and supportive treatment is prolonged, with palliative care being basically provided. Quality of life then appears as an essential challenge to be reached by patients, family members and health professionals. According to the World Health Organization, quality of life refers to the individual's perception of their position in life, in the context of the culture and value system in which they live, and in relation to their goals, expectations, standards and concerns. In addition, there is the concept of "health-related quality of life", which assesses the impact of health on the individual's ability to live fully. Thus, the health/disease process of people with SCA is governed by hereditary, biological and environmental factors and also suffers interference from the social environment, gender, race/ethnicity and class inequalities, which consequently compromise the factors considered acquired.

In patients with SCA, physical, emotional and social changes cause losses in quality of life. These changes result from the various complications that can arise over the natural course of the disease, in addition to the decrease in the life expectancy of the individual. SCA causes limitations in the lives of patients, with pain and several hospitalizations, most likely, responsible for the physical and emotional destabilization of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell anemia, of both sexes, aged ≥ 18 years.
* Patients who have clinical stability and are eligible for the treatment protocol.

Exclusion Criteria:

* Presence of comorbidities not related to sickle cell anemia.
* Patients with inability to perform the six-minute walk test.
* Patients who have cognitive impairment that impairs their inclusion in the study.
* Abandonment of treatment during the application of the protocol.
* Uncontrolled hypertension or use of psychotropic drugs.
* Any significant limitations due to osteoarthropathy.
* Have had any orthopedic surgery in the previous year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-07-25 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life related to activities of daily living through the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) before and after the execution of the treatment plan. | 12 weeks
  The SF-36 is composed of 11 questions and 36 items that comprise eight components (domains or dimensions), represented by functional capacity (10 items), physical aspects (four items), pain (two items), general health status (five items), vitality (four items), social aspects (two items), emotional aspects (three items), mental health (five items) and a comparative question about the current perception of health for a year. The individual receives a score in each domain, which ranges from 0 to 100, with 0 being the worst score and 100 being the best (PIMENTA et. Al, 2008).

SECONDARY OUTCOMES:
Peripheral muscle function before and after the execution of the treatment plan. | 12 weeks
  The peripheral muscle function will be evaluated through handgrip strength (HGS) and quadriceps strength (QS). HGS will be measured by a maximal isometric strength test with the SH5001 device (Saehan Corporation, Korea) in the dominant upper limb. The participants will be positioned according to standard recommendations, with their elbow flexed at 90°, the forearm half-pronated, and the wrist in a neutral position. HGS was summarized as the highest value of three attempts with a 60-s rest time. The QS will be evaluated with a tension dynamometer (sensor capacity = 200 kg, E-lastic 5.0, E-sports SE, Brazil). The range of motion within 90° during the test will be determined, starting at 90° flexion at the knee. The maximum force will be assessed in the dominant leg after a 5-s sustained isometric contraction. QS will be summarized as the highest value from three attempts with a 1-min intervals.
Functional capacity through the 6-minute walk test (6MWT) before and after the execution of the treatment plan. | 12 weeks
  The 6MWT will be performed according to previously described recommendations using a 30-m runway demarcated with cones at both ends. Blood pressure, heart rate, respiratory rate, peripheral oxygen saturation, and Borg's perceived exertion scale will be measured before and after the 6MWT.

CONTACTS AND LOCATIONS:
Overall Officials: Agnaldo J Lopes, PhD, Principal Investigator — Centro Universitário Augusto Motta
Locations (1):
- Agnaldo José Lopes, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Almeida A, Roberts I. Bone involvement in sickle cell disease. Br J Haematol. 2005 May;129(4):482-90. doi: 10.1111/j.1365-2141.2005.05476.x. PMID 15877730
- [Result] Baltich J, Emery CA, Stefanyshyn D, Nigg BM. The effects of isolated ankle strengthening and functional balance training on strength, running mechanics, postural control and injury prevention in novice runners: design of a randomized controlled trial. BMC Musculoskelet Disord. 2014 Dec 4;15:407. doi: 10.1186/1471-2474-15-407. PMID 25471989
- [Result] Chatel B, Hourde C, Gondin J, Foure A, Le Fur Y, Vilmen C, Bernard M, Messonnier LA, Bendahan D. Impaired muscle force production and higher fatigability in a mouse model of sickle cell disease. Blood Cells Mol Dis. 2017 Mar;63:37-44. doi: 10.1016/j.bcmd.2017.01.004. Epub 2017 Jan 11. PMID 28110136
- [Result] Chaturvedi S, DeBaun MR. Evolution of sickle cell disease from a life-threatening disease of children to a chronic disease of adults: The last 40 years. Am J Hematol. 2016 Jan;91(1):5-14. doi: 10.1002/ajh.24235. PMID 26547630
- [Result] Dougherty KA, Schall JI, Rovner AJ, Stallings VA, Zemel BS. Attenuated maximal muscle strength and peak power in children with sickle cell disease. J Pediatr Hematol Oncol. 2011 Mar;33(2):93-7. doi: 10.1097/MPH.0b013e318200ef49. PMID 21228717
- [Result] Maioli MC, Soares AR, Bedirian R, Alves UD, de Lima Marinho C, Lopes AJ. Relationship between pulmonary and cardiac abnormalities in sickle cell disease: implications for the management of patients. Rev Bras Hematol Hemoter. 2016 Jan-Feb;38(1):21-7. doi: 10.1016/j.bjhh.2015.11.001. Epub 2015 Dec 11. PMID 26969771
- [Result] Milner PF, Kraus AP, Sebes JI, Sleeper LA, Dukes KA, Embury SH, Bellevue R, Koshy M, Moohr JW, Smith J. Sickle cell disease as a cause of osteonecrosis of the femoral head. N Engl J Med. 1991 Nov 21;325(21):1476-81. doi: 10.1056/NEJM199111213252104. PMID 1944426
- [Result] Ohara DG, Ruas G, Walsh IA, Castro SS, Jamami M. Lung function and six-minute walk test performance in individuals with sickle cell disease. Braz J Phys Ther. 2014 Jan-Feb;18(1):79-87. doi: 10.1590/s1413-35552012005000139. PMID 24675916
- [Result] Piel FB, Patil AP, Howes RE, Nyangiri OA, Gething PW, Dewi M, Temperley WH, Williams TN, Weatherall DJ, Hay SI. Global epidemiology of sickle haemoglobin in neonates: a contemporary geostatistical model-based map and population estimates. Lancet. 2013 Jan 12;381(9861):142-51. doi: 10.1016/S0140-6736(12)61229-X. Epub 2012 Oct 25. PMID 23103089
- [Result] Ravelojaona M, Feasson L, Oyono-Enguelle S, Vincent L, Djoubairou B, Ewa'Sama Essoue C, Messonnier LA. Evidence for a profound remodeling of skeletal muscle and its microvasculature in sickle cell anemia. Am J Pathol. 2015 May;185(5):1448-56. doi: 10.1016/j.ajpath.2015.01.023. Epub 2015 Mar 13. PMID 25773175
- [Result] Rubio MA, Diez L, Alvarez N, Munteis E. [Muscle involvement in sickle cell disease]. Med Clin (Barc). 2015 Nov 6;145(9):413-4. doi: 10.1016/j.medcli.2014.12.010. Epub 2015 Feb 7. No abstract available. Spanish. PMID 25662725
- [Derived] Almeida CHS, Reis LFDF, Nascimento LPADS, Soares AR, Maioli MCP, Lopes AJ. Therapist-oriented home rehabilitation for adults with sickle cell anemia: effects on muscle strength, functional capacity, and quality of life. Hematology. 2021 Dec;26(1):612-619. doi: 10.1080/16078454.2021.1965736. PMID 34411499